CLINICAL TRIAL: NCT02683551
Title: Comparison of Effects of Energy Based Devices on Quality of Life After Sutureless Thyroidectomy?
Brief Title: Comparison of QoL for Sutureless Thyroidectomy
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Akif Enes ARIKAN, MD, Istanbul University
Other Study IDs: IUCTF-EndSx-2015-01; 83045809/604.01/02 (Other: Ethical Committee)
Record Dates: First submitted 2015-10-24; First posted 2016-02-17 (Estimated); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Thyroidectomy; Quality of Life

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Ligasure: Patients underwent to Sutureless Thyroidectomy with Ligasure SmallJaw
  Interventions: Procedure: Sutureless Thyroidectomy
- Harmonic: Patients underwent to Sutureless Thyroidectomy with Harmonic FOCUS
  Interventions: Procedure: Sutureless Thyroidectomy

INTERVENTIONS:
Procedure: Sutureless Thyroidectomy — Thyroidectomy performed with energy based devices and no use of ligation. Used device is not altered for this study. Non of the personnel in the operating room including surgical team knows if the patient was enrolled or not in this study.

SUMMARY:
Patients underwent thyroidectomy filled an computer or paper based QoL questionnaire before and after operation.

DETAILED DESCRIPTION:
Patients who have consent to undergo to total thyroidectomy with sutureless technique (regardless of attending to study or not) for benign thyroid diseases in the institution are asked to participate to this study. Patients are informed that participating to this study will not alter their treatment method. Patients were operated either with Ligasure SmallJaw or Harmonic Focus according to result of label picked from bag. Same surgical team performed all operations and they did not know if the patient was participated in study or not.

Patients willing to participate in this study are being questioned for their quality of life (QoL) with a patient-reported outcome (PRO) questionnaire before surgery and 4 weeks after surgery. For assessment of quality of life Thy-PRO-39 questionnaire is being used. Responses of patients to QoL questionnaire is being recorded to a secure online database. After data completion answers of patients will be exported as anonymous to principal investigator for analysis. Effect of two energy based devices (EBD) on QOL will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Sutureless thyroidectomy for benign conditions

Exclusion Criteria:

* Known neck malignity,
* History of neck operation
* Ligation use during surgery
* Refusal of patient
* Non-capable patient
* Non-euthyroid patient
* Pregnancy
* Having rheumatic diseases
* Having connective tissue diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who has planned to undergo to sutureless thyroidectomy for benign conditions.
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Overall alterations in quality of life according to Thy-PRO-39 questionnaire | 4 weeks

SECONDARY OUTCOMES:
Alterations in social life according to Thy-PRO-39 questionnaire | 4 weeks
Alterations in daily life according to Thy-PRO-39 questionnaire | 4 weeks
Alterations in Tiredness according to Thy-PRO-39 questionnaire | 4 weeks
Alterations in cognitive complaints according to Thy-PRO-39 questionnaire | 4 weeks
Alterations in anxiety according to Thy-PRO-39 questionnaire | 4 weeks
Alterations in depressivity according to Thy-PRO-39 questionnaire | 4 weeks
Alterations in emotional susceptibility according to Thy-PRO-39 questionnaire | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ates OZYEGIN, Prof, MD, Study Director — Istanbul University, Cerrahpasa Medical Faculty

REFERENCES:
- [Background] Watt T, Bjorner JB, Groenvold M, Cramon P, Winther KH, Hegedus L, Bonnema SJ, Rasmussen AK, Ware JE Jr, Feldt-Rasmussen U. Development of a Short Version of the Thyroid-Related Patient-Reported Outcome ThyPRO. Thyroid. 2015 Oct;25(10):1069-79. doi: 10.1089/thy.2015.0209. Epub 2015 Aug 26. PMID 26214034
- See also: Data collection and information release system — http://www.drenes.com/